CLINICAL TRIAL: NCT03204214
Title: Binge Drinking And Addiction : Case-Control Study in Hospital
Acronym: BACH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marie-Pierre TAVOLACCI (Other)
Responsible Party: Sponsor-Investigator, Marie-Pierre TAVOLACCI, Doctor, University Hospital, Rouen
Organization: University Hospital, Rouen (Other)
Other Study IDs: 2016/166/OB
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Alcohol Dependence
Keywords: binge drinking
MeSH Terms: conditions — Alcoholism; Binge Drinking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Case Control Study :

Objective:

Frequent Binge drinking during 18-25 years is a risk factor of alcohol addiction in adulthood (25-40 years) Hypothesis: 25% of frequent binge drinking, OR = 2, power 80%, alpha risk : 5% 126 Cases aged 25 to 40 years: alcohol addict patients recruited in Addiction Unit in Rouen University Hospital 126 controls aged 25 to 40 years: non alcohol addict recruited by the Clinical investigation center in Rouen University Hospital An anonymous self-questionnaire was completed Binge Drinking during 18-25 years was retrospectively evaluated Confusion biais was also recorded

ELIGIBILITY:
Inclusion Criteria

* 25 to 40 years:
* alcohol addiction for the cases

Exclusion criteria

* age <20 and >40
* alcohol addiction for the controls

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases recruited in Addiction Unit in Rouen University Hospital Controls recruited by the Clinical investigation center in Rouen University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Frequent binge drinking | 18-25 years old

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre TAVOLACCI, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tavolacci MP, Berthon Q, Cerasuolo D, Dechelotte P, Ladner J, Baguet A. Does binge drinking between the age of 18 and 25 years predict alcohol dependence in adulthood? A retrospective case-control study in France. BMJ Open. 2019 May 5;9(5):e026375. doi: 10.1136/bmjopen-2018-026375. PMID 31061035